CLINICAL TRIAL: NCT01384825
Title: Observational Study of the Prevalence of CCSVI in Multiple Sclerosis and in Other Neurodegenerative Diseases
Acronym: COSMO
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: FISM 2010R1
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis; Neurodegenerative Diseases
Keywords: Multiple Sclerosis; Other Neurodegenerative Diseases; Chronic CerebroSpinal Venous Insufficiency; Prevalence; Case-control
MeSH Terms: conditions — Multiple Sclerosis; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MS: Subjects with Multiple Sclerosis
- HC: Healthy Controls
- OND: Subjects with Other Neurodegenerative Diseases, including both other non-inflammatory neurodegenerative diseases ("OND") and other inflammatory neurodegenerative diseases ("ONDi")

SUMMARY:
The presence of abnormalities in the cerebral venous circulation, defined as Chronic Cerebrospinal Venous Insufficiency (CCSVI), has recently been reported in patients with Multiple Sclerosis (MS), in healthy subjects and in subjects with other neurological diseases. These reports have aroused much interest both in the scientific world and, above all, among the communities of patients and Associations having the aim of aiding people with MS and of promoting scientific research into this disease.

In the literature published so far there is a lack of verification in large samples of the prevalence of CCSVI in MS compared with that observed in healthy subjects and in those with other diseases of the nervous system.

This is an observational study investigating the prevalence of CCSVI in subjects with MS and comparing it with the prevalence observed in a control population consisting of Healthy Controls (HC) and in a population affected by other neurological diseases of the central nervous system of degenerative, vascular, inflammatory and autoimmune origin.

A total of at least 1,200 adults with MS will be included in the study, as well as 400 healthy subjects and 400 subjects with other neurodegenerative diseases.

DETAILED DESCRIPTION:
It has been recently reported the possible presence of abnormalities in the cerebral venous circulation of people with MS, in healthy controls and in people with other neurological diseases. These reports have aroused much interest both in the scientific world and, above all, among the communities of patients and Associations having the aim of aiding people with MS and of promoting scientific research into this disease. In particular, the studies by Zamboni and colleagues (Ferrara University) and by Zivadinov and colleagues (University of Buffalo) have suggested an association between CCSVI and MS that was widely reported by the mass media world-wide.

It can be noted that in the literature published so far there is a lack of verification in large samples of the prevalence of CCSVI in MS compared with that observed in healthy subjects and in those with other diseases of the nervous system. The recent and authoritative contributions from the scientific community involved with MS stressing the need for closely controlled and suitably designed clinical studies for investigating the hypotheses suggested with regard to CCSVI (with the necessary thoroughness and with the promptness demanded by the public opinion) are therefore definitely justified.

The possibility that there may be a new pathogenic mechanism underlying the development of MS, not in line with the majority of the experimental data concerning the aetiopathogenesis of this disease, has produced a strong echo throughout the scientific community. Increasingly, in recent months, both the working groups mentioned above and new authors have developed further research studies in order to confirm and extend the results obtained and to lay scientifically sound foundations for possible therapeutic applications for this discovery.

The Fondazione Italiana Sclerosi Multipla (FISM) Onlus, in its capacity as Promoter of this study, wishes, responsibly, to produce the best possible answer for people with MS all over the world. It therefore feels that it is necessary to proceed with the utmost scientific thoroughness, initially by means of a large-scale sample study for evaluating the prevalence of venous abnormalities in MS compared with that observed in normal controls and in controls with other diseases of the nervous system. In this context, the features of this study that distinguish it from previous studies and from the current state of knowledge are the following:

1. Blind multi-Site observational study using the Echo-Color-Doppler equipment assigned to the study;
2. Size of the sample with MS, of at least 1200 study subjects;
3. Evaluation of the prevalence of CCSVI and of other malformations of the venous haemodynamics in the Clinically Isolated Syndrome (CIS), Relapsing-Remitting (RR), Primary Progressive (PP) and Secondary Progressive (SP) forms of MS, using a larger sample than those involved up to the present time.

In this observational study, the prevalence of CCSVI and of other malformations of the venous haemodynamics will be evaluated in different forms of MS and in other diseases of the nervous system. This is therefore an observational study investigating the prevalence of CCSVI in subjects with MS and comparing it with the prevalence observed in a control population consisting of healthy subjects and in a population of people with other neurological diseases of the central and peripheral nervous system of degenerative, vascular, inflammatory and autoimmune origin.

The study is a multi-Site observational study. A total of at least 1,200 adults with MS will be included in the study, as well as 400 healthy subjects and 400 subjects with other neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

Group A (MS)

* Age: 18 to 55;
* Subjects of either sex with a diagnosis of MS according to McDonald's criteria and subsequent revisions (38, 39) and patients with CIS;
* Course of the disease: RR - SP - PP - CIS;
* Duration of the disease: from 1 month to 25 years for RR, SP and PP subjects; 5 years at most for the subjects with CIS,
* Not in a period of clinical relapsing of the disease (at least 30 days since the last clinical relapse),
* Subjects treated or not with immunomodulating and immunosuppressive drugs;
* Signature of the informed consent form.

Group B (HC)

* Age: 18 to 55;
* No significant diseases and no familiarity for MS, that is to say healthy controls (HC);
* Signature of the informed consent form. The subjects included in this group may be, for instance, non-blood relatives or spouses of the subjects with MS or with any of the other diseases being studied, or be linked to them by ties of affinity (e.g. a son-in-law with a father-in-law, a husband with his wife's brother, etc.) or accompanying persons or operators from other Sites.

Group C (OND)

* Age: 18 to 55 ;
* Subjects with other non-inflammatory neurodegenerative diseases (OND) such as, by way of example, Parkinson's disease, amyotrophic lateral sclerosis (ALS) and heredoataxia.
* Signature of the informed consent form.

Group D (ONDi)

* Age: 18 - 55
* Patients with other inflammatory neurodegenerative diseases (ONDi) such as, by way of example, optical neuromyelitis (ONM), acute disseminated encephalomyelitis (ADEM), encephalitis, neurolupus, neurological complications of systemic autoimmune diseases.
* Signature of the informed consent form.

Exclusion Criteria:

* Presence of acute or chronic diseases of an invalidating nature or that could interfere with the design and aims of the study;
* Clinically ascertained heart disease (New YOrk Heart AssoCiation (NYHA) Class ≥ I).
* Past episodes of venous thromboembolism (including both Deep Vein Thrombosis and lung embolism).
* Tumours.
* Thrombophilia as defined in the case history.
* Diabetes.
* Primitive or secondary pulmonary hypertension and related treatment.
* Concomitant systemic steroid treatment or in the last 30 days.
* Current or past cerebrovascular disease.
* Episodes of Transient Global Amnesia (TGA).
* Obvious pregnancy.
* Past diagnosis of CCSVI or earlier treatment for CCSVI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of at least 1,200 adults with MS will be included in the study, as well as 400 healthy subjects and 400 subjects with other neurodegenerative diseases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of CCSVI | The primary outcome will be assessed at enrollment (day 1). No follow-up is planned.
  The prevalence of CCSVI in MS (overall and in its various different forms) will be estimated, with 95% confidence intervals, and compared with that of the other groups. The differences in the prevalence of CCSVI between the various groups will be evaluated using the chi-square test. The sensitivity, specificity and accuracy of the method will be estimated with their 95% confidence intervals. Values of p equal to or lower than 0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni L Mancardi, MD, Principal Investigator — Università di Genova - Dipartimento di Neuroscienze, Oftalmologia e Genetica - Via De Toni, 5 - Genova; Giancarlo Comi, Principal Investigator — Divisione di Neurologia e Servizio di Neurofisiologia, Ospedale San Raffaele di Milano
Locations (43):
- Italy (42):
  - Azienda Ospedali Riuniti - Div. di Neurologia - Centro Studi Sclerosi Multipla, Ancona
  - Università di Bari - Ospedale Consorziale Policlinico - Dip. Scienze Neurologiche e Psichiatriche, Bari
  - Azienda USL Città di Bologna - Distretto Santo Stefano Savena - Centro Sclerosi Multipla, Bologna
  - Azienda Ospedaliera Spedali Civili Presidio Montichiari - Centro Studi Sclerosi Multipla, Brescia
  - Università degli Studi di Cagliari - Centro Sclerosi Multipla - Ospedale Binaghi, Cagliari
  - Azienda Ospedaliera "Garibaldi" - U.O. Neurologia, Catania
  - Azienda Ospedaliera Universitaria "Policlinico Vittorio Emanuele" - Istituto Scienze Neurologiche, Catania
  - Istituto San Raffaele Giuseppe Giglio - Centro Sclerosi Multipla, Cefalù
  - Ospedale Universitario G. D'Annunzio - Centro Sclerosi Multipla, Chieti
  - Azienda Ospedaliera San Giuseppe - Centro Scl. Multipla - U.O. Neurologia, Empoli
  - Università degli Studi di Ferrara Arcispedale Sant'Anna - Clinica Neurologica, Ferrara
  - Università degli Studi di Ferrara Arcispedale Sant'Anna - Istituto di Clinica Neurologica, Ferrara
  - Azienda Ospedaliero Universitaria Careggi - Centro di Riferimento Regionale per la Sclerosi Multipla, Florence
  - Azienda Ospedaliero Universitaria Careggi - Centro Sclerosi Multipla, Florence
  - Azienda Ospedaliera Universitaria Ospedali Riuniti - Centro Sclerosi Multipla, Foggia
  - Ospedale S. Antonio Abate - Centro Studi Sclerosi Multipla, Gallarate
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Ospedale S. Andrea - Divisione di Neurologia, La Spezia
  - Ospedale Tappeiner - Div. Neurologica, Merano
  - IRCCS Centro Studi Neurolesi "Bonino Pulejo" di Messina, Messina
  - Azienda Ospedaliera Universitaria "G. Martino" - Dipartimento Neuroscienze Psichiatria e Anestesiologia, Messina
  - Università degli Studi di Milano - Dipartimento di Neurologia - Ospedale S. Raffaele - Via Olgettina , 60, Milan
  - Fondazione Ist. Neurologico Besta - Centro Sclerosi Multipla, Milan
  - Fondazione Don Carlo Gnocchi, IRCCS Santa Maria Nascente - Unità Operativa Sclerosi Multipla, Milan
  - Ospedale Niguarda Cà Granda - Centro Sclerosi Multipla, Milan
  - Università Federico II - Clinica Neurologica II, Napoli
  - Azienda Ospedaliera S. Luigi - Centro Sclerosi Multipla - Divisione Universitaria di Neurologia, Orbassano
  - Policlinico Az. Ospedaliera - Clinica Neurologica I, Padua
  - Università degli Studi di Palermo - Istituto di Neuropsichiatria - A.O.U.P. "P. Giaccone", Palermo
  - Azienda Ospedaliera Villa Sofia C.T.O. - Neurologia Padiglione Geriatrico, Palermo
  - Istituto Neurologico C. Mondino - Divisione di Neurologia, Pavia
  - Arciospedale S. Maria Nuova - Centro Studi Sclerosi Multipla, Reggio Emilia
  - Università Tor Vergata - Clinica Neurologica - Dipartimento di Neuroscienze, Roma
  - Ospedale Sant'Andrea - Neurologia e Centro Neurologico Terapie Sperimentali, Roma
  - Università di Sassari - Clinica Neurologica, Sassari
  - Università degli Studi di Siena - Dip. di Neuroscienze - Sez. Neurologia, Siena
  - Università degli Studi di Siena - Dip. di Neuroscienze - U.O. Neurologia e Malattie Neurometaboliche, Siena
  - Azienda Ospedaliera Universitaria S. Giovanni Battista - Centro Sclerosi Multipla - Dipartimento di Neuroscienze, Torino
  - Azienda Ospedaliera "Ca Foncello" - Dipartimento di Neuroscienze - U.O. Neurologia, Treviso
  - Ospedale di Cattinara - Istituto Clinica Neurologica, Trieste
  - Ospedale S. Bortolo - Divisione di Neurologia - Centro Sclerosi Multipla, Vicenza
  - Azienda Sanitaria Provinciale di Ragusa Ospedale "R. Guzzardi" - U.O.C. Neurologia e Neurofisiopatologia, Stroke Unit, Vittoria
- Opera Contract Research Organization SRL, Timișoara, Timiș County, Romania